CLINICAL TRIAL: NCT00371982
Title: Effect of Fish Oil on Adiposity and Atherogenic Factors in Type 2 Diabetic Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INSERM-237-6900, Paris 6-069
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2002-11

CONDITIONS: Type 2 Diabetes
Keywords: Fish oil; Type 2 diabetic women; adiposity; adipose tissue inflammation; PAI-1; Insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Insulin Resistance | interventions — Fish Oils; Maxepa

INTERVENTIONS:
Drug: Fish oil (Maxepa)

SUMMARY:
1. whether the intake of n-3 PUFA has additional effects on insulin sensitivity and adiposity (total fat mass and adipocyte morphology and function) in T2D women.
2. n-3 PUFA supplementation might influence inflammatory genes expression in the adipose tissue of T2D patients.

DETAILED DESCRIPTION:
Thus, the present study was designed to evaluate the effects of n-3 PUFAs dietary supplementation on lipid and glucose homeostasis and to address the impact of this treatment on adiposity and adipose tissue gene expression in T2D women.A total of 27 T2D women (BMI 27-35kg/m², age 40-60 y) were randomly allocated to two months of 3 g/day of either fish oil (1.8 g n-3 PUFA) or placebo (paraffin oil), in a double-blind parallel design.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic postmenopausal women
2. glycaemia of 7.87-14.0 mmol/l, HbA1c of 7 to 10.5%
3. plasma triglycerides between 1.72-4.6 mmol/l,
4. aged between 40 -60,
5. BMI: 27-40 kg/m2
6. able to swallow tablets

Exclusion Criteria:

1. patients with abnormal renal, hepatic and thyroid functions as determined by physical examination, blood cell count and standard blood biochemical profile
2. patients with gastrointestinal disorders
3. patients treated with thiazolidinediones or insulin

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2002-12; Study Completion 2005-04

PRIMARY OUTCOMES:
The effect of 2 month treatment on:
adiposity (total fat mass, adipocyte morphology), atherogenic markers and insulin sensitivity

SECONDARY OUTCOMES:
the underlying mechanisms of the observed results and tried to define new targets of fish oil metabolic effects
and the impact of fish oil on systemic inflammatory markers and adipose tissue inflammatory genes.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa W Rizkalla, MD,PhD, Study Director — INSERM (National institution of Health and Medical Research); Gerard Slama, MD, professor, Study Chair — Public Assistance-Paris Hospitals (AP-HP), University Paris 6
Locations (1):
- Department of Diabetes-Hotel Dieu Hospital, Paris, France